CLINICAL TRIAL: NCT06565403
Title: Treatment of Critically Ill Patients With Acute Kidney Injury and Dialysis in the Intensive Care Unit
Brief Title: Hyperlactatemia in Critically Ill Patients With Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Collaborators: University of Maribor, Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, Robert Ekart, Prof.Robert Ekart, MD, PhD, University Medical Centre Maribor
Other Study IDs: UMC Maribor
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; lactate; acidosis; survival
MeSH Terms: conditions — Acute Kidney Injury; Acidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the research is to determine the prevalence of patients with acute kidney injury in the intensive care unit, the role of dialysis treatment in the treatment of these patients.

DETAILED DESCRIPTION:
A retrospective and observational study was conducted in which the investigators included participants who were hospitalised in the Department of Internal Intensive Care Medicine at the University Hospital Maribor and who required replacement haemodialysis treatment during their hospital stay. The decision on haemodialysis treatment was made after an agreement between the attending specialist in intensive care medicine and the nephrologist if there was a clear indication for starting replacement haemodialysis treatment. It should be emphasised that each of the patients received an appropriate form of treatment according to indication and clinical condition, in line with all relevant recommendations and guidelines.

The investigators collected data on the underlying comorbidities, the indication for ICU treatment, the indication for starting haemodialysis treatment, the type of haemodialysis (continuous venovenous haemodialysis, continuous venovenous haemodiafiltration) and the basic parameters of haemodialysis (level of ultrafiltration and total ultrafiltration, anticoagulants used, duration of procedures, complications during haemodialysis, prescribed and achieved haemodialysis dose with emphasis on the amount of dialysate/substitute/ultrafiltrate used (Qe, effluent dose), number of haemodialysis procedures, dialysis membrane used with or without immunoadsorbent membrane). The investigators collected data on laboratory results (haemoglobin, leucocytes, platelets, C-reactive protein, procalcitonin, lactate, urea, creatinine, bilirubin, albumin, partial pressure of oxygen in arterial blood, myoglobin, lactate dehydrogenase, Interleukin-6, beta-2-microglobulin, cystatin C), some measured haemodynamic/vital parameters (mean arterial pressure, diuresis, oxygen demand) and the dose of vasopressor drugs during treatment. The investigators analysed all the data obtained and attempted to objectively evaluate the success of the treatment. The investigators compared different haemodialysis membranes (standard membranes for continuous haemodialysis vs. newer membranes such as Emic-2® and Oxiris membrane®), different dialysis techniques (haemodialysis vs. haemodiafiltration) and the effects of using the Cytosorb® immunoadsorptive membrane. The investigators have obtained data on the duration of hospitalisation and survival of participants after treatment (up to 1 year).

We analysed the data using basic statistical methods, where a value of p < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* presence of acute kidney injury, stage 3 according to Kidney Disease:Improving Global Outcomes (KDIGO) criteria
* treatment with renal replacement therapy (RRT)

Exclusion Criteria:

* patients with chronic kidney disease (CKD) receiving chronic RRT
* previous known malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All critically ill patients with stage 3 AKI who received RRT were included in the final study cohort.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Hyperlactatemia in critically ill patients with acute kidney injury treated with renal replacement therapy in the intensive care unit | 90 days
  survival

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Ekart, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make statistical data analysis available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year.
Access Criteria: The member of the research team.

REFERENCES:
- [Derived] Ekart R, Kobal B, Korosec T, Jakopin E, Svensek F, Piko N, Bevc S, Hojs R. Hyperlactatemia in critically ill patients with acute kidney injury treated with renal replacement therapy in the intensive care unit. BMC Nephrol. 2025 Apr 30;26(1):217. doi: 10.1186/s12882-025-04149-5. PMID 40307699